CLINICAL TRIAL: NCT02665117
Title: Preventing Metabolic Side Effects of Thiazide Diuretics With KMgCitrate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Wanpen Vongpatanasin, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STU 092015-058
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Results first posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Hypertension
Keywords: Hypokalemia; Isoprostanes; Insulin resistance; Aldosterone; Hepatic fat; Muscle Magnesium; Liver fat
MeSH Terms: conditions — Hypertension; Hypokalemia; Insulin Resistance; Fatty Liver | interventions — potassium-magnesium citrate; Potassium, Dietary; Chlorthalidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KMgCit + Chlorthalidone (Active Comparator): After a run-in period of 2-3 weeks on Chlorthalidone, patients will be randomized to the addition of KMgCit for 4 months.
  Interventions: Drug: Potassium Magnesium Citrate (KMgCit); Drug: Chlorthalidone
- KCl + Chlorthalidone (Active Comparator): After a run-in period of 2-3 weeks on Chlorthalidone, patients will be randomized to the addition of KCl for 4 months.
  Interventions: Drug: Potassium Chloride (KCl); Drug: Chlorthalidone

INTERVENTIONS:
Drug: Potassium Magnesium Citrate (KMgCit) — KMgCit will be administer for 4 months with chlorthalidone.
  Other Names: KMgCit
  Arms: KMgCit + Chlorthalidone
Drug: Potassium Chloride (KCl) — KCl will be administer for 4 months with chlorthalidone.
  Other Names: KCl
  Arms: KCl + Chlorthalidone
Drug: Chlorthalidone — Chlorthalidone will be administered for 2-3 weeks. Then either KCL or KMgCit will be added to Chlorthalidone and the combination will be taken for 4 months.

SUMMARY:
Chlorthalidone (CTD) may produce various metabolic disturbances, including hypokalemia, activation of Renin-Angiotensin- Aldosterone (RAA) system, oxidative stress, dyslipidemia, Fibroblast growth factor 23 (FGF23) synthesis, and magnesium depletion. These factors may interact with each other to contribute to the development of insulin resistances and metabolic syndrome. Smaller studies have suggested that Potassium magnesium Citrate (KMgCit) can ameliorate CTD- induced metabolic side effects independent of correction of hypokalemia. This study will tests if KMgCit ameliorates CTD induced metabolic effects independent of correction of hypokalemia.

DETAILED DESCRIPTION:
CTD- induced metabolic side effects were though to be dependent on hypokalemia, but subsequent studies suggested that CTD - induced side effects were independent from hypokalemia. On the other hand, magnesium depletion has been linked to increased Renin-Angiotensin- Aldosterone (RAA) system, the development of metabolic syndrome and insulin resistance with magnesium supplementation ameliorating these effects.

Participants will participate in a double-blinded, parallel design study. After baseline evaluation participants will take Chlorthalidone (CTD) alone for 2-3 weeks. They will then be randomized to two equal groups to take KMgCit powder or Potassium Chloride (KCl) powder along with CTD for 4 months.

We speculate that Mg depletion is responsible for hepatic fat deposition, which then produces insulin resistance. Co-administration of KMgCit powder would avert magnesium (Mg) depletion, block hepatic fat deposition by restoring normal Mg status and direct intestinal binding of fat, thereby ameliorating insulin resistance. To test this hypothesis, we shall quantitate muscle Mg status and hepatic fat content by magnetic resonance spectroscopy (MRS) before and after KMgCit. Change in fasting glucose, insulin resistance, serum potassium, FGF23, and aldosterone will be compared between KCL and KMgCit groups after 4 months.

ELIGIBILITY:
Inclusion Criteria:

• Treated or untreated stage I hypertension

Exclusion Criteria:

* Diabetes mellitus,
* Renal impairment (serum creatinine > 1.4 mg/dL),
* Any heart diseases such as congestive heart failure, sustained arrhythmia, or coronary heart disease,
* Chronic regular NSAID use,
* Allergy to thiazide diuretics,
* Gastro-esophageal reflux disease (GERD) requiring treatment with acid reducing agents or antacid more than once a week,
* Esophageal-gastric ulcer or history of gastrointestinal bleeding,
* Chronic diarrhea, vomiting,
* Excessive sweating,
* Unprovoked hypokalemia (serum K < 3.5 mmol/L) or hyperkalemia (serum K > 5.3 mmol/L),
* Abnormal liver function test (Aspartate transaminase (AST) or Alanine transaminase (ALT) above upper limit of normal range),
* Subjects on any potassium supplement on a regular basis for any reason, such as patients with primary aldosteronism,
* Pregnancy,
* History of major depression, bipolar disorder, or schizophrenia,
* History of substance abuse,
* Gout,
* Metabolic alkalosis, with serum bicarbonate > 32 meq/L,
* Severe dietary salt restriction, less than1/2 spoonful or 50 meq sodium/day.
* Patient with Claustrophobia will not have MRI but can still participate in the study without MRI
* Metal implants will not have MRI but can still participate in the study without MRI

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-01; Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wanpen Vongpatanasin, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (3):
- United States (3):
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Background] Ahmed LA. Protective effects of magnesium supplementation on metabolic energy derangements in lipopolysaccharide-induced cardiotoxicity in mice. Eur J Pharmacol. 2012 Nov 5;694(1-3):75-81. doi: 10.1016/j.ejphar.2012.07.036. Epub 2012 Aug 23. PMID 22939974
- [Background] Carter BL, Einhorn PT, Brands M, He J, Cutler JA, Whelton PK, Bakris GL, Brancati FL, Cushman WC, Oparil S, Wright JT Jr; Working Group from the National Heart, Lung, and Blood Institute. Thiazide-induced dysglycemia: call for research from a working group from the national heart, lung, and blood institute. Hypertension. 2008 Jul;52(1):30-6. doi: 10.1161/HYPERTENSIONAHA.108.114389. Epub 2008 May 26. No abstract available. PMID 18504319
- [Background] Guerrero-Romero F, Rodriguez-Moran M. Hypomagnesemia, oxidative stress, inflammation, and metabolic syndrome. Diabetes Metab Res Rev. 2006 Nov-Dec;22(6):471-6. doi: 10.1002/dmrr.644. PMID 16598698
- [Background] Hata A, Doi Y, Ninomiya T, Mukai N, Hirakawa Y, Hata J, Ozawa M, Uchida K, Shirota T, Kitazono T, Kiyohara Y. Magnesium intake decreases Type 2 diabetes risk through the improvement of insulin resistance and inflammation: the Hisayama Study. Diabet Med. 2013 Dec;30(12):1487-94. doi: 10.1111/dme.12250. Epub 2013 Jun 29. PMID 23758216
- [Background] Koenig K, Padalino P, Alexandrides G, Pak CY. Bioavailability of potassium and magnesium, and citraturic response from potassium-magnesium citrate. J Urol. 1991 Feb;145(2):330-4. doi: 10.1016/s0022-5347(17)38330-1. PMID 1988724
- [Background] Odvina CV, Mason RP, Pak CY. Prevention of thiazide-induced hypokalemia without magnesium depletion by potassium-magnesium-citrate. Am J Ther. 2006 Mar-Apr;13(2):101-8. doi: 10.1097/01.mjt.0000149922.16098.c0. PMID 16645424
- [Background] Pak CY. Correction of thiazide-induced hypomagnesemia by potassium-magnesium citrate from review of prior trials. Clin Nephrol. 2000 Oct;54(4):271-5. PMID 11076102
- [Background] Price AL, Lingvay I, Szczepaniak EW, Wiebel J, Victor RG, Szczepaniak LS. The metabolic cost of lowering blood pressure with hydrochlorothiazide. Diabetol Metab Syndr. 2013 Jul 9;5(1):35. doi: 10.1186/1758-5996-5-35. PMID 23837919
- [Background] Ruml LA, Pak CY. Effect of potassium magnesium citrate on thiazide-induced hypokalemia and magnesium loss. Am J Kidney Dis. 1999 Jul;34(1):107-13. doi: 10.1016/s0272-6386(99)70115-0. PMID 10401023
- [Derived] Vongpatanasin W, Giacona JM, Pittman D, Murillo A, Khan G, Wang J, Johnson T, Ren J, Moe OW, Pak CCY. Potassium Magnesium Citrate Is Superior to Potassium Chloride in Reversing Metabolic Side Effects of Chlorthalidone. Hypertension. 2023 Dec;80(12):2611-2620. doi: 10.1161/HYPERTENSIONAHA.123.21932. Epub 2023 Oct 17. PMID 37846572

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | KMgCit + Chlorthalidone | KCl + Chlorthalidone
Started | 30 | 31
Completed | 29 | 31
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KMgCit + Chlorthalidone | KCl + Chlorthalidone | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (9.3) | 58.1 (12.8) | 59.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 15 | 20 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 26 | 29 | 55
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Fasting Plasma Glucose From Week 4 to Week 16
Description: Fasting plasma glucose was measured from venous blood sample at week 4 and week 16
Time Frame: week 4 and week 16
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | KMgCit + Chlorthalidone | KCl + Chlorthalidone
Number analyzed (Participants) | 29 | 31
mg/dL | -5.6 (13.3) | 2.3 (9.9)

2. Secondary Outcome: Chang in Hepatic Fat Measured at Baseline and Week 16
Description: Will be measured using hepatic magnetic resonance imaging at baseline and at week 16
Time Frame: baseline to week 16
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | KMgCit + Chlorthalidone | KCl + Chlorthalidone
Number analyzed (Participants) | 19 | 19
percent | 0.31 (2.74) | 1.59 (4.9)

3. Secondary Outcome: Change in Muscle Magnesium Content Measured at Baseline and Week 16
Description: Will be measured using magnetic resonance imaging at baseline and at week 16
Time Frame: baseline to week 16
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | KMgCit + Chlorthalidone | KCl + Chlorthalidone
Number analyzed (Participants) | 19 | 19
mM | -0.01 (0.1) | 0.02 (0.08)

4. Secondary Outcome: Change in FGF23 From Week 4 to Week 16
Description: Will be measured from venous blood sample from week 4 to week 16
Time Frame: week 4 to week 16
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | KMgCit + Chlorthalidone | KCl + Chlorthalidone
Number analyzed (Participants) | 29 | 31
pg/ml | 38.1 (123.3) | 13.6 (104.1)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | KMgCit + Chlorthalidone | KCl + Chlorthalidone
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 2/29 | 0/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KMgCit + Chlorthalidone (N=29) | KCl + Chlorthalidone (N=31)
Mechanical Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — mechanical tibia/fibula fracture
Syncopal Episode (General disorders) | 1 (1) | 0 (0) — Syncopal episode in clinic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-08-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT02665117/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT02665117/ICF_001.pdf